CLINICAL TRIAL: NCT04858958
Title: A Phase Ib, Randomized, Open-label, Multi-center Study to Evaluate the Preliminary Efficacy and Safety of Furmonertinib Mesilate in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer Harboring EGFR Exon 20 Insertion Mutation
Brief Title: Study of FURMONERTINIB in Patients With NSCLC Having Exon 20 Insertion Mutation
Acronym: FAVOUR
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol No.: ALSC012AST2818
Record Dates: First submitted 2021-04-12; First posted 2021-04-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- treated subjects will receive Furmonertinib 160mg/day, (Experimental): treated subjects will receive Furmonertinib 160mg/day, QD, PO, under fasted state, until progressive disease, death or intolerability.
  Interventions: Drug: Furmonertinib 160mg
- treated subjects will receive Furmonertinib 240mg/day, (Experimental): treated subjects will receive Furmonertinib 160mg/day, QD, PO, under fasted state, until progressive disease, death or intolerability.
  Interventions: Drug: Furmonertinib 240mg
- treatment-naïve subjects will receive Furmonertinib 240mg/day (Experimental): Treatment naïve patients with EGFR exon 20 insertion mutation positive NSCLC
  Interventions: Drug: Furmonertinib 240mg

INTERVENTIONS:
Drug: Furmonertinib 160mg — randomized to 160mg QD
  Arms: treated subjects will receive Furmonertinib 160mg/day,
Drug: Furmonertinib 240mg — randomized to 240mg QD
  Arms: treated subjects will receive Furmonertinib 240mg/day,; treatment-naïve subjects will receive Furmonertinib 240mg/day

SUMMARY:
This is a phase Ⅰb multi-center clinical study. To explore the preliminary efficacy and safety of Furmonertinib Mesilate at different doses in locally advanced or metastatic NSCLC patients with EGFR exon 20 insertion mutation.

The study plans to enroll 30 subjects, including 20 treated patients and 10 treatment-naïve patients. The subjects with disease progression after previous systematic anti-tumor therapy will be randomized to receive Furmonertinib Mesilate 160 mg/day (N=10) or 240 mg/day (N=10), respectively. The treatment-naïve patients do not need to be randomized and all will receive Furmonertinib Mesilate 240 mg/day (N=10) until disease progression, death or intolerability.

The primary endpoint is ORR; the secondary study endpoints include DCR, DOR, DepOR, PFS, OS, CNS ORR, safety and the PK profile of Furmonertinib Mesilate and its metabolites (AST5902).

In addition, the peripheral blood ctDNA will be collected and analyzed in this study

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥18 years;
* Histologically or cytopathologically confirmed primary non-small cell lung cancer (NSCLC) with predominant non-squamous cell histology;
* The treated patients must have radiological disease progression following the last anti-tumor therapy; and the treatment-naïve patients must have documented positive EGFR exon 20 insertion mutation by laboratory tests prior to enrollment;
* Subjects meeting either of the following conditions (in accordance with the AJCC 8th edition TNM stage classification for lung cancer):
* Treated patients: patients with locally advanced (judged by investigators as not suitable for surgery or radiotherapy) or metastatic NSCLC who are confirmed to have radiological or pathological disease progression during or after the last systematic anti-tumor therapy before the first dose of investigational product
* Treatment-naïve patients: patients with locally advanced (judged by investigators as not suitable for surgery or radiotherapy) or metastatic NSCLC who have no prior systematic anti-tumor therapy before the first dose of investigational product. If the time from the completion of adjuvant or neoadjuvant therapy to the first disease progression is > 6 months, the patients will be eligible for enrollment to the study; if it is ≤6 months, the patients will be regarded as treated patients and evaluated in accordance with the criteria for treated patients
* Having at least one measurable lesion (in accordance with RECIST1.1). Note: measurable lesion can neither be subject to local therapy as radiotherapy nor used for biopsy in screening period; if there is only one measurable lesion, this lesion will be permitted to be biopsied. However, the baseline radiological examination can be performed for this lesion at least 14 days after biopsy.
* Adequate organ function as shown in the laboratory test, including:
* Life expectancy >12 weeks after the first dose of investigational product;
* Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of investigational product; female subjects of non-childbearing potential may not undergo pregnancy test or contraception. Non-childbearing potential is defined as: 50 years and above, no use of hormone therapy and amenorrhea for at least 12 months; or having received sterilization operation. Female subjects at childbearing age and male subjects agree to take effective contraceptive measures during the study and within 6 months after drug discontinuation;
* Being able to understand and voluntarily participate in the study, and sign the informed consent form.

Exclusion Criteria:

* NSCLC with predominant squamous cell histology, small cell lung cancer or neuroendocrine carcinoma indicated by Histology or cytology test;
* Expected to receive other anti-tumor therapy other than the investigational product during the study;
* Treatment-naïve patients: having previously received systematic anti-tumor therapy targeting EGFR pathway (marketed drugs or drugs under development, EGFR TKI or antibody)
* Treated patients: having previously received systematic anti-tumor therapy with 3rd-generation EGFR TKI (marketed drugs or drugs under development) ;
* Having received the following therapies:
* Having been irradiated for >30% bone marrow or a large area within 4 weeks prior to the first dose of investigational product;
* Having received major surgery within 4 weeks prior to the first dose of investigational product or plan to receive major surgery during the study with exception of the surgical procedures to establish vascular access, biopsy through mediastinoscopy or thoracoscopy;
* Use of a potent CYP3A4 inhibitor within 7 days prior to the first dose of investigational product or a potent CYP3A4 inducer within 21 days prior to the first dose of investigational product; use of the traditional Chinese medicine or traditional Chinese medicine preparation with tumor indication, or traditional Chinese medicine or traditional Chinese medicine preparation with adjuvant anti-tumor effect within two weeks prior to the first dose of investigational product or expected to be required during the study;
* Having participated in the clinical trial and received the investigational product or device within 4 weeks or at least 5 half-lives prior to the first dose of investigational product;
* Having received other anti-tumor drugs within 14 days prior to the first dose of investigational product;
* Concurrent spinal cord compression or symptomatic brain metastasis. Subjects with stable brain metastasis will be eligible. Stable brain metastasis is defined as the patients who have completed regular treatment for brain metastasis, are clinically stable or asymptomatic for at least two weeks and do not need steroid therapy. If the investigator considers there is no indication of immediate radical treatment, patients with asymptomatic brain metastasis will be eligible.
* The toxicity caused by previous anti-tumor therapy has not recovered to ≤CTCAE grade 1 (CTCAE 5.0) ( except alopecia, sequelae of previous platinum-related neurotoxicity) or the level specified in the inclusion/exclusion criteria;
* Unstable pleural effusion or peritoneal effusion with obvious symptoms; those with stable clinical symptoms for at least 28 days after drainage of pleural effusion or ascites will be eligible;
* Having a history of other malignant tumor, or other concurrent malignant tumors (except those that have undergone radical operation and have no recurrence within 5 years post operation, e.g., cervical carcinoma in situ, basal cell carcinoma of skin and papillary thyroid carcinoma);
* Previous interstitial lung disease (ILD), drug-induced interstitial lung disease, radiation pneumonitis requiring steroid therapy; or having the clinical manifestations of suspected interstitial lung disease;
* Having severe or uncontrolled systemic disease requiring treatment that is considered by investigators as ineligible for the study, including hypertension, diabetes, chronic heart failure (NYHA Functional Classification III-IV), unstable angina pectoris, myocardial infarction within one year, active hemorrhagic disease, etc.;
* Left ventricular ejection fraction (LVEF) <50% on echocardiography;
* Clinically significant prolonged QT interval or other arrhythmia or clinical status considered by investigators that may increase the risk of prolonged QT interval; for example, QTc>470 ms on ECG at resting state, complete left bundle branch block, degree III atrioventricular block, congenital long QT syndrome, serious hypokalemia, or current use of drugs that may lead to prolonged QT interval;
* Serious gastrointestinal dysfunction, or disease that may affect the intake, transportation or absorption of investigational product;
* Known hepatitis B virus (positive HBsAg), hepatitis C virus (positive HCV Ab) or human immunodeficiency virus (positive HIV antibody) infection;
* Infectious disease requiring intravenous medication;
* Known history of mental disease or drug abuse, and currently having an attack or still taking drugs;
* Known or suspected allergy to Furmonertinib or other components of its preparation;
* Female subjects or female partners of male subjects who are pregnant or lactating, or plan to be pregnant during the study;
* Poor compliance, inability to comply with the study procedures, restriction or requirements;
* Other conditions that are considered by investigators as unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
ORR, objective response rate | up to 12 months
  The proportion of subjects who achieve Complete Response (CR) and Partial Response (PR) by the best response from the first dose of Furmonertinib to the end of study.

SECONDARY OUTCOMES:
DCR, | up to 12 months
  The proportion of subjects who achieve CR, PR, and Stable Disease (SD) by the best response from the first dose of Furmonertinib to the end of study.
DOR | up to 12 months
  The proportion of subjects who achieve CR, PR, and Stable Disease (SD) by the best response from the first dose of Furmonertinib to the end of study.
PFS | up to 12 months
  PFS is defined as the time from randomization or start of study treatment until objective tumor progression or death depending on study protocol

CONTACTS AND LOCATIONS:
Overall Officials: Baohui C Han, PHd, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided